CLINICAL TRIAL: NCT04013958
Title: Comparison of Treatment by IM Ketamine to IV Ketamine in Patients With Renal Colic
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director, R&D Department, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TASMC-19-DT-0060-19-CTIL
Record Dates: First submitted 2019-07-07; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Acute Pain; Renal Colic
Keywords: Morphine; Ketamine; Renal colic
MeSH Terms: conditions — Acute Pain; Renal Colic | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized according to a blocked randomization scheme "WWW.RANDOMIZATION.COM" , which permits assignment of the participant to either group "A" or "group B" (the IM ketamine+IV morphine group or IV ketamine+IV morphine with IM saline (placebo) group.
  Eligible patients will be divided in equal proportions (50 in group A and 50 in group B).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV Ketamine (Active Comparator): IV Ketamine group will receive IV Ketamine with IV morphine and IM saline.
  Interventions: Drug: IV Ketamine
- IM Ketamine (Experimental): IM Ketamine group will receive IM Ketamine with IV morphine.
  Interventions: Drug: IM Ketamine

INTERVENTIONS:
Drug: IV Ketamine — IV Ketamine 0.1 mg/kg with IV morphine -0.1 mg/kg with IM Sailne 0.9%
  Other Names: No other
  Arms: IV Ketamine
Drug: IM Ketamine — IM Ketamine 0.3 mg/kg with IV morphine -0.1 mg/kg
  Arms: IM Ketamine

SUMMARY:
Patients who present to the emergency department (ED), with acute pain due to renal colic, are often treated with opioids. Treatment with opioids has many disadvantages - cardio-respiratory depression, nausea, vomiting and long term dependence. For these reasons, there is a constant search for a way to reduce the use of opioids. ketamine has been proven to augmented the analgesic effect of opioids, and thus reduce the use and adverse effects of opioids. Different studies about the use of Ketamine as a sedition agent have shown that Ketamine given IM versus IV has longer duration of effect with less adverse effects.

The study we are conducting is designed to test and analyze the safety and efficacy of IV Ketamine with IV Morphine compared to IV Ketamine and morphine with IM placebo in a setting of acute pain due to, or suspected renal colic in the ED. When both ways of administration are given by the protocol as is customary for treatment of pain in the Emergency Medicine department, and will be a prospective, randomized, double blind, controlled study.

DETAILED DESCRIPTION:
The procedure:

1. Eligible patients will be identified by the ED personnel.
2. Research physician will address the patient, explain about the trial and ask the patient to sign a consent form.
3. The patient will be randomized and assigned to a trial group: "A" or "B" and it will be noted in the Data sheet.
4. According to physician order (IV amount and IM amount) and patient group assignment, the nurse will prepare and administer the different drugs.
5. Patients in group "A" wiil receive IV Ketamine with IV morphine and IM placebo of normal saline. Patients in group "B" wiil receive IM Ketamine with IV morphine.
6. The amount will be calculated based on the patients' weight:

   IV Morphine -0.1 mg/kg: Morphine vial contains 10 mg/10 ml. IV Ketamine -0.1 mg/kg: Ketamine vial contains 50 mg/1 ml. IM Ketamine -0.25 mg/kg: Ketamine vial contains 50 mg/1 ml.
7. Prior to administering medication to the patient a research assistant, who is blinded to the choice of drugs given, will measure vital signs (blood pressure, heart rate and O2 saturation) as well as pain level on a 100 mm VAS (visual analogue scale) questionnaire.
8. After administration of medications the researcher assistant will measure vital signs (blood pressure, heart rate and O2 saturation) as well as pain level on a 100 mm VAS questionnaire, at 5 and 10 minutes after administration, and then at 30, 45, 60, and 90 minutes.
9. Measurement of vital signs will not interfere with any other treatment that the patients receives for their injury in the ED.
10. Cardiorespiratory follow-up (as per bullet point number 8 above), will be concluded at 1.5 hours post-intervention, and clinical follow-up will continue as long as the patient remains in the ED.
11. During the time of the the followup and after, if pain had not subsided sufficiently according to treating physician's clinical assessment, patient will receive further analgesic medications by physician order, as per ED protocol. The protocol takes into account concurrent medications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Self-report pain greater than or equal to 7/10 on a numerical-verbal scale
* Weigh 50-100 kg
* Have systolic blood pressure of 90-180 mmHg
* Have an ASA (American Society of Anaesthesiologists' classification) score of 1-2

Exclusion Criteria:

* Have had opioid analgesia administered within 6 hours of the study
* Are chronic analgesia users (of opioid or others)
* Have known allergies to morphine or ketamine
* Are pregnant
* Have a psychiatric history

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of IM Ketamine in decreasing pain intensity [patient assessed - VAS pain score] | 1.5 hour post administration
  Time to achieve a clinically meaningful pain reduction was defined as the first time-point at which the patient reported 15mm of pain reduction or more. Maximal pain reduction was defined as the lowest VAS score reported by the patient over the course of follow-up. Time to maximal pain reduction was defined as the time at which the patient has the lowest VAS score over the course of the 1.5 hours follow-up.
Adverse effects [Opiate Related Symptom Distress Scale] | 1.5 hour post administration
  adverse effects [Opiate Related Symptom Distress Scale] [ Time Frame: 1.5 hour post administration ]

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, department of Emergency Medicine, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
a table summering pain assessing questioners will be available from corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP